CLINICAL TRIAL: NCT02954328
Title: The Effect of Transcranial Direct Current Stimulation (tDCS) on Motor and Cognitive Functions in Idiopathic Fallers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director of Research and Development, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-16-NG-0699-CTIL
Record Dates: First submitted 2016-10-31; First posted 2016-11-03 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Elderly Idiopathic Fallers
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tDCS (Experimental): The active tDCS condition will consist of 4 visit:
  During each visit, subject will receive a single 20-minute session targeting the prefrontal cortices of either real (1.5 mA) or sham tDCS. Total 4 different targets:
  1. Sham
  2. motor M1 area
  3. motor M1 + Dorsolateral Prefrontal cortex
  4. Dorsolateral Prefrontal cortex.
  The tDCS condition will be randomized and double blinded
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — The active tDCS condition will consist of 20 min of continuous stimulation. This amount of stimulation is safe for healthy young and older adults and has been shown to induce acute beneficial changes in cortical excitability and cognitive functions.
  Other Names: Transcranial Direct Current Stimulation

SUMMARY:
The concurrent performance of two tasks, i.e., dual tasking (DT), is a common and ubiquitous every day phenomena. For example, people frequently walk while talking on a cellphone or drive while talking to a passenger. Often, the performance of one or more of these simultaneously performed tasks may deteriorate when another task is carried out at the same time, even in healthy young adults. This reduction in performance is referred to as the DT deficit or DT cost and is typically much higher in Idiopathic Fallers (IF) than in age-matched controls. In this population the DT cost impairs the gait pattern, as manifested, for example, in increased gait variability, exacerbating instability and fall risk.

In the proposed study, would be evaluated the effects of tDCS on dual tasking performance following tDCS.

The researchers expect that stimulation of the Pre Frontal Cortex (PFC) (using tDCS) will increase DT performance and prefrontal activation.

DETAILED DESCRIPTION:
tDCS intervention: Noninvasive tDCS will be delivered by study personnel uninvolved with any other study procedures. In the study will be used a battery-driven electrical stimulator. Stimulation and sham condition will be performed based on previous studies. Briefly, the anode will be placed over the PFC and the cathode over the right supraorbital region. The real tDCS condition will consist of 20 min of continuous stimulation at target intensity of 1.5 mA. This amount of stimulation is safe for healthy young and older adults and has been shown to induce acute beneficial changes in cortical excitability and cognitive functions. For the sham condition, an inactive stimulation protocol would be followed, as compared with an 'off-target' active protocol, in order to minimize participant risk.

Pre- and post-tDCS assessments will include:

Gait assessment: Gait parameters will include both spatial and temporal parameters obtained using body fixed wearable sensors (accelerometers and gyroscopes) [Weiss et al. 2015; Ben et al. 2015]. Parameters will include (but are not limited to) gait speed, stride length and stride time as well as rhythmicity measures such as stride to stride variability and gait regularity.

Fall history and fear of falling will also be assessed (e.g., Falls Efficacy Scale International, FES-I) to further characterize the cohort and explore possible confounds.

Cognitive assessment: A detailed computerized cognitive battery that has been used extensively at TASMC in different cohorts [Dwolatzky et al. 2003;Hausdorff et al. 2006;Springer et al. 2006;Yogev et al. 2005;Aarsland et al. 2003] will quantify several cognitive domains including working memory, executive function, verbal function, problem solving, a global cognitive score, and attention.

ELIGIBILITY:
Inclusion Criteria:

1. age 65-85 years,
2. ability to walk for 6 minutes unassisted,
3. adequate vision capabilities, and
4. stable medications for the past month.

Exclusion Criteria:

1. diagnosis of stroke, Parkinson's disease, peripheral neuropathy or other neurologic disorder,
2. lower-extremity deformity, joint replacement, severe arthritis or other diagnosed musculoskeletal disorder that may influence gait,
3. orthostatic hypotension, recent history of syncope or vertigo,
4. myocardial infarction or surgery within the past 6 months,
5. any unstable medical condition,
6. psychiatric co-morbidity (e.g., major depressive disorder as determined by DSM V criteria),
7. likely dementia (i.e., Mini Mental State Exam score < 24 or based on DSM V),
8. sedating medications (sedatives, anti-psychotics, hypnotics, anti-depressants,
9. colorblindness (confounder for cognitive assessment), or
10. contraindications to tDCS

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Immediate change in gait speed | 1st measure will be taken at baseline ans 2nd immediate post intervention
  Gait speed will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance.

SECONDARY OUTCOMES:
fNIRS related frontal lobe activation - changes in tissue oxygenation | 1st measure will be taken at baseline ans 2nd immediate post intervention
  fNIRS will be used to investigate the role of the frontal lobe in DT walking and how it is affected by tDCS.The fNIR system provides with real-time monitoring of tissue oxygenation in the brain as subjects take different tests.
Changes in cognitive performance - Executive Function composite score | 1st measure will be taken at baseline ans 2nd immediate post intervention
  The NeuroTrax software uses tests of cognitive performance that measure similar cognitive functions to traditional paper-based tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, Prof., Principal Investigator — Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
Locations (2):
- Hebrew Rehabilitation Center / Harvard Medical School, Roslindale, Massachusetts, United States
- Laboratory for Gait and Neurodynamics, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou J, Hao Y, Wang Y, Jor'dan A, Pascual-Leone A, Zhang J, Fang J, Manor B. Transcranial direct current stimulation reduces the cost of performing a cognitive task on gait and postural control. Eur J Neurosci. 2014 Apr;39(8):1343-8. doi: 10.1111/ejn.12492. Epub 2014 Jan 20. PMID 24443958
- [Derived] Schneider N, Dagan M, Katz R, Thumm PC, Brozgol M, Giladi N, Manor B, Mirelman A, Hausdorff JM. Combining transcranial direct current stimulation with a motor-cognitive task: the impact on dual-task walking costs in older adults. J Neuroeng Rehabil. 2021 Feb 1;18(1):23. doi: 10.1186/s12984-021-00826-2. PMID 33526043